CLINICAL TRIAL: NCT04233112
Title: Assessing the Efficacy of Melatonin and Osteogenic Loading on Bone Health in an Osteopenic Population: MelaOstrong Study
Brief Title: Melatonin and Osteogenic Loading on Osteopenia
Acronym: MelaOstrong
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: OsteoStrong (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/08/15
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Melatonin; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Placebo/Mock (Placebo Comparator): Placebo capsules; mock osteogenic loading
  Interventions: Device: Mock for Osteogenic Loading; Drug: Placebo (plant fiber) for melatonin
- Melatonin/Mock (Experimental): Melatonin capsules; mock osteogenic loading
  Interventions: Drug: Melatonin 5 mg; Device: Mock for Osteogenic Loading
- Placebo/Osteogenic loading (Experimental): Placebo capsules/osteogenic loading
  Interventions: Device: Osteogenic loading; Drug: Placebo (plant fiber) for melatonin
- Melatonin/Osteogenic loading (Experimental): Melatonin capsules/osteogenic loading
  Interventions: Drug: Melatonin 5 mg; Device: Osteogenic loading

INTERVENTIONS:
Drug: Melatonin 5 mg — Capsules containing 5mg melatonin will be prepared by Delta Care RX™ Pharmacy. Participants will be asked to take them nightly for one year.
  Arms: Melatonin/Mock; Melatonin/Osteogenic loading
Device: Osteogenic loading — Osteogenic loading device therapy includes the emulation of impact forces through kinetic chains of natural impact absorption with fixtures that have the ability to capture bone compression data. Participants will be asked to perform osteogenic loading once per week.
  Arms: Melatonin/Osteogenic loading; Placebo/Osteogenic loading
Device: Mock for Osteogenic Loading — Mock osteogenic loading will occur using the osteogenic loading device therapy includes the emulation of impact forces through kinetic chains of natural impact absorption with fixtures that have the ability to capture bone compression data. Participants will be asked to perform mock osteogenic loading once per week.
  Arms: Melatonin/Mock; Placebo/Mock
Drug: Placebo (plant fiber) for melatonin — Capsules containing plant fiber will be prepared by Delta Care RX™ Pharmacy. Participants will be asked to take them nightly for one year.
  Arms: Placebo/Mock; Placebo/Osteogenic loading

SUMMARY:
This study will be assessing the efficacy of melatonin and/or osteogenic loading on modulating bone health in an osteopenic population.

ELIGIBILITY:
Inclusion criteria: To be included in the study, the participant must be a male or female with osteopenia (T-score between -1.0 and -2.5) who is at least 18 years of age. The participant must be willing to undergo an osteogenic loading protocol once per week and/or take a pill (placebo or melatonin) for one year. The participant must also be willing to come to the study location to receive their monthly capsules and to provide urine, have their blood pressure taken and complete questionnaires on 3 occasions (baseline/month 0, month 3 and month 12). The study participants must also be willing to get a DXA scan at months 0 and 12 at one of the three Weinstein Imaging locations.

Exclusion criteria: Women or men with osteoporosis; women or men with osteopenia due to hyperparathyroidism, multiple myeloma, metastatic bone disease, chronic steroid use including corticosteroids; women or men who are on any bone therapies (i.e. bisphosphonates, selective estrogen receptor modulators (SERMs), hormone therapy, teriparatide, and denosumab); men and women with chronic obstructive pulmonary disease (COPD); women or men who smoke; pregnant women; and men or women with muscular dystrophy, unmedicated hypertension, or unrepaired hernia, restrictions to movement and exercise, and parathyroid dysfunctions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | O-12 months
  Bone mineral density (BMD) at baseline (month 0) and month 12. Bone density will be assessed by dual energy x-ray absorptiometry (DXA) scan at baseline (month 0) and at month 12. Bone density, expressed as percentage change from baseline (T-scores), will be compared within and between groups at 12 mos.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Witt-Enderby, PhD, Principal Investigator — Duquesne University
Locations (2):
- United States (2):
  - OsteoStrong® in Scott Towne Center, Pittsburgh, Pennsylvania
  - Duquesne University, Pittsburgh, Pennsylvania